CLINICAL TRIAL: NCT07399769
Title: Efficacy and Safety of MSLN CAR-T in Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen University General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 112
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Malignant Tumors (With Positive Expression of MSLN in Tumor Tissue)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CART group (Experimental): Participants will receive lymphodepleting chemotherapy (FC regimen: Fludarabine + Cyclophosphamide) on Days -5, -4, and
  -3 relative to the planned MSLN CAR-T cell infusion. The CAR-T cell infusion will be administered 72 hours after the completion of the FC chemotherapy.
  Interventions: Combination Product: CAR-T

INTERVENTIONS:
Combination Product: CAR-T — Participants will receive lymphodepleting chemotherapy (FC regimen: Fludarabine + Cyclophosphamide) on Days -5, -4, and
  -3 relative to the planned MSLN CAR-T cell infusion. The CAR-T cell infusion will be administered 72 hours after the completion of the FC chemotherapy.

SUMMARY:
1. Study Title:

   Efficacy and safety of MSLN CAR-T in advanced malignant tumors
2. Study Objectives:

   Primary: To evaluate the safety and tolerability of MSLN-targeted CAR-T cell therapy in patients with stage III/IV advanced malignant tumors.

   Secondary: To preliminarily evaluate the efficacy of MSLN-targeted CAR-T cell therapy in this patient population.

   Exploratory: To assess in vivo expansion and persistence of infused MSLN-targeted CAR-T cells and explore correlations with clinical outcomes.
3. Participant Intervention:

Participants will receive lymphodepleting chemotherapy (FC regimen: Fludarabine + Cyclophosphamide) on Days -5, -4, and

-3 relative to the planned MSLN CAR-T cell infusion. The CAR-T cell infusion will be administered 72 hours after the completion of the FC chemotherapy.

DETAILED DESCRIPTION:
Detailed Description:

This is a prospective, interventional Phase I/II clinical study designed to evaluate the safety and efficacy of MSLN-targeted CAR-T cell therapy in patients with advanced malignant tumors. A total of 20 patients aged 18-75 years with unresectable, locally advanced, recurrent, or metastatic solid malignancies will be enrolled. All patients must have histopathologically confirmed disease and positive MSLN expression in tumor tissue.

MSLN CAR-T cells will be administered as a single intravenous infusion at a total dose of 0.5-2 × 10^6 CAR-T cells/kg. Eligible subjects (N=20) will be assigned by the investigator to receive MSLN CAR-T cell infusion.

Endpoints:

* Primary Endpoint:

  o Incidence and severity of treatment-emergent adverse events (TEAEs) within 30 days after MSLN CAR-T cell infusion.
* Secondary Endpoints:

  * Objective response rate (ORR = CR + PR) assessed within 8 weeks after infusion;
  * Overall survival (OS) and progression-free survival (PFS) at 6 months;
  * In vivo expansion and persistence kinetics of infused CAR-T cells.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years (≥18 and ≤75 years), either sex;
2. The subject voluntarily participates in the study and provides written informed consent signed by the subject or his/her legally authorized representative;
3. Histopathologically confirmed unresectable, locally advanced, recurrent, or metastatic solid malignant tumor; according to the AJCC TNM staging system (8th edition, 2017), subjects diagnosed with stage III or stage IV solid malignant tumors;
4. Presence of measurable and evaluable lesions according to RECIST v1.1;
5. Positive MSLN expression in tumor tissue confirmed by immunohistochemistry (IHC);
6. The subject must have received standard first-line therapy and has experienced disease progression or is intolerant to such therapy;
7. The subject is not suitable for curative treatment modalities such as definitive chemoradiotherapy and/or surgery/immune checkpoint inhibitors, or refuses surgical resection;
8. No antibody-based therapy administered within 2 weeks prior to cell therapy;
9. ECOG performance status 0-2;
10. No contraindications to peripheral blood leukapheresis;
11. Estimated life expectancy ≥ 3 months.

Exclusion Criteria:

1. History of allergy to any component of the cell product;
2. Any of the following hematologic abnormalities on complete blood count (CBC): WBC ≤ 1 × 10^9/L, absolute neutrophil count (ANC) ≤ 0.5 × 10^9/L, absolute lymphocyte count (ALC) ≤ 0.5 × 10^9/L, or platelets (PLT) ≤ 25 × 10^9/L;
3. Any of the following laboratory abnormalities, including but not limited to: serum total bilirubin ≥ 1.5 mg/dL; serum ALT or AST > 2.5 × ULN; serum creatinine ≥ 2.0 mg/dL;
4. NYHA class III or IV heart failure per the New York Heart Association functional classification, or left ventricular ejection fraction (LVEF) < 50% on echocardiography;
5. Abnormal pulmonary function with oxygen saturation (SpO₂) < 92% on room air;
6. History of myocardial infarction, coronary angioplasty or stenting, unstable angina, or other clinically significant severe cardiac disease within 12 months prior to enrollment;
7. Grade 3 hypertension with poor blood pressure control despite medical treatment;
8. History of traumatic brain injury, disturbance of consciousness, epilepsy, or severe cerebral ischemic or hemorrhagic disease;
9. Presence of autoimmune disease, immunodeficiency, or other conditions requiring immunosuppressive therapy;
10. Presence of uncontrolled active infection;
11. Prior treatment with any CAR-T cell product or other genetically modified T-cell therapy;
12. Receipt of a live vaccine within 4 weeks prior to enrollment;
13. Positive test results for HIV, HBV, HCV, and TPPA/RPR, and/or HBV carriers;
14. History of alcohol abuse, illicit drug use, or psychiatric disorders;
15. Participation in any other clinical study within 3 months prior to enrollment;
16. Female subjects meeting any of the following:

    1. pregnant or breastfeeding; or
    2. planning pregnancy during the study period; or
    3. of childbearing potential and unable/unwilling to use effective contraception;
17. Any other condition that, in the opinion of the investigator, makes the subject unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
TRAEs | From date of initial treatment to the 30 days after treatment
  Adverse events during treatment

SECONDARY OUTCOMES:
Disease-related clinical responses | From date of enrollment until the date of clinical responses,up to 2 years
  Disease-related clinical responses include CR/PR/SD/PD

CONTACTS AND LOCATIONS:
Overall Officials: Li Yu, Principal Investigator — Shenzhen University General Hospital
Locations (1):
- Shenzhen University General Hospital, Shenzhen, Other (Non U.s.), China

IPD SHARING:
Plan to Share IPD: No